CLINICAL TRIAL: NCT06623864
Title: Significant Activities in the Implementation of the Integrated Person-centered Care Model: Intervention Protocol
Brief Title: Significant Activities in the Integrated Person-centered Care Model
Acronym: IO/20240924
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Burgos (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: IO/20240924
Record Dates: First submitted 2024-09-24; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Old Age; Dementia; Old Age; Debility
MeSH Terms: conditions — Alzheimer Disease; Frailty

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- single group (Experimental): The intervention proposal will be developed in a module with 10 elderly people, all of them men, with moderate dependence and older, with an average age of 84 years. All of them have multiple medical pathologies with the need for continuous nursing care.
  Interventions: Other: meaningful activities
- CONTROL GROUP (Experimental): The intervention proposal will be developed in a module with 10 elderly people, all of them men, with moderate dependence and older, with an average age of 84 years. All of them have multiple medical pathologies with the need for continuous nursing care.
  Interventions: Other: other activities

INTERVENTIONS:
Other: meaningful activities — The intervention proposal will be developed in a module with 27 elderly people, all of them men, with moderate dependence and older, with an average age of 84 years. All of them have multiple medical pathologies with the need for continuous nursing care.
  Arms: single group
Other: other activities — The intervention proposal will be developed in a module with 27 elderly people, all of them men, with moderate dependence and older, with an average age of 84 years. All of them have multiple medical pathologies with the need for continuous nursing care.
  Arms: CONTROL GROUP

SUMMARY:
The increasing life expectancy and global aging population necessitate changes in long-term gerontological services based on Person-Centred Care approaches. This study aims to improve Person-Centred Care in geriatric centers through meaningful activities and the role of occupational therapists and direct care professionals in developing these activities. A descriptive cross-sectional quasi-experimental design was proposed, with 10 participants.

DETAILED DESCRIPTION:
Background: Increasing life expectancy means that the ageing of populations globally is on the rise. It is therefore important to promote changes in long-term gerontological services based on Person-Centred Care approaches, in which meaningful occupation serves as a basis and is supported by appropriate professional support, such as the occupational therapist and the direct care professional.

Objective: To improve Person-Centred Care in a geriatric centre, through the use of meaningful activities and to identify the role of the occupational therapist and direct care professional in the development of these activities.

Methods: A descriptive cross-sectional quasi-experimental pre-post single-group design is proposed. A total of 10 participants. The methodology used will be mixed. The data collection techniques and tools will be the PDC evaluation instrument pre and post intervention and a survey at the end of the project.

ELIGIBILITY:
Inclusion Criteria:

* That the direct care worker has a degree as a nursing assistant, dependency care technician, geroculturist or certificate of professionalism.
* The worker must speak and understand Spanish.
* The residence must offer service during the day, in the morning or afternoon shift.
* Workers must have been with the department for more than 4 months.

Exclusion Criteria:

* Workers who work night shift only.
* Workers on rotating shifts in all departments of the residence.
* Workers absent at the time of the study due to temporary leave, vacations or other causes.

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Kruskal-Wallis test | 3 months
  To compare the medians of the groups
Spearman's correlation coefficient | 3 months
  This measure allows us to determine the strength and direction of the association between the variables

CONTACTS AND LOCATIONS:
Locations (1):
- Olalla Saiz Vazquez, Burgos, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No
Although each participant will provide their name and email address to register for the study, their data and survey results will be completely anonymous and linked to a participant code. On each measurement occasion, participants will be emailed a link to the survey and, when clicked, will be taken to the google-forms web platform that will host the surveys. The web surveys will not ask for any information that can be used to identify a specific participant, and google-forms will not record any metadata.

REFERENCES:
- [Background] McCormack, B., & McCance, T. (2017). Person-Centred Practice in Nursing and Health Care: Theory and Practice. Wiley-Blackwell.
- [Background] World Health Organization. (2016). Framework on Integrated, People-Centred Health Services. WHO.
- [Background] Gittell, J. H., & Vidal, M. (2018). Relational Coordination: Guidelines for Theory and Practice. Oxford University Press.
- [Background] Edvardsson, D., & Innes, A. (2017). Measuring Person-Centred Care: A Review of Tools and Methodologies. Journal of Nursing Scholarship, 49(2), 223-235. https://doi.org/10.1111/jnu.12276
- [Background] Dewing, J. (2008). Person-Centred Dementia Care: A Vision to Be Realised. Journal of Nursing Management, 16(3), 261-268. https://doi.org/10.1111/j.1365-2834.2007.00848.x